CLINICAL TRIAL: NCT05531539
Title: 2nd Clinical Trial of WELMO System With Respiratory Patients
Brief Title: Evaluation of Wearable Vest for Lung Monitoring
Acronym: WELMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: George Papanicolaou Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WELMO-THESS
Record Dates: First submitted 2022-08-22; First posted 2022-09-08 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Chronic Lung Disease
Keywords: respiratory disease; lung auscultation; Electric Impedance Tomography; sensors; biosignals acquisition
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Outpatient Respiratory patients (Experimental): They were examined with spirometry, manual auscultation of the thorax and where necessary, with chest X-ray or CT scan. They wore the WELMO sensors vest for a period of 15-20 minutes during which they performed tidal and deep breathing, cough and spirometry maneuvers and changes of posture. At the end of the study, they were requested to fill in a questionnaire about comfort and usability of the vest.
  Interventions: Device: WELMO sensors vest
- Hospitalized Respiratory patients (Experimental): They were examined with spirometry, manual auscultation of the thorax and where necessary, with chest X-ray or CT scan. They wore the WELMO sensors vest for a period of 15-20 minutes during which they performed tidal and deep breathing, cough and spirometry maneuvers and changes of posture. At the end of the study, they were requested to fill in a questionnaire about comfort and usability of the vest.
  Interventions: Device: WELMO sensors vest
- Critically ill Respiratory patients (Experimental): They were examined with manual auscultation of the thorax and where necessary, with chest X-ray or CT scan. They wore the WELMO sensors vest for a period of 15-20 minutes during which the vest recorded the breathing provided by the mechanical ventilator.
  Interventions: Device: WELMO sensors vest

INTERVENTIONS:
Device: WELMO sensors vest — Wearing of a vest equipped with lung auscultation and EIT sensors for signal acquisition and transmission

SUMMARY:
This was the pilot study of the EU funded research and innovation project WELMO (Wearable Electronics for Effective Lung Monitoring) -Grant agreement number: 825572. The clinical trial involved patients suffering from a variety of respiratory pathological conditions and examined the ease-of-use and efficacy of the WELMO system, comprising a sensors vest for thorax auscultation and recording of Electric Impedance Tomography (EIT) signals and transmitting those on the cloud for review by physicians. The study recruited and briefly monitored 27 patients who underwent brief training and subsequent wearing of the sensors vest for 15-20 minutes, after manual auscultation, spirometry and oximetry. The collected data were transmitted wirelessly to a tablet and then securely to the cloud for review by attending physicians. The usability of the system, the quality of the obtained signals and the validity of the results were evaluated.

DETAILED DESCRIPTION:
The study recruited and briefly monitored 27 patients at the outpatient department and the medical ward of the Pulmonology Department of "G. Papanikolaou" General Hospital of Thessaloniki, Greece, as well as the 1st Intensive Care Unit of the same Hospital. Patients were recruited during their hospitalization or at the outpatient setting and informed consent was obtained before participation. They were examined with spirometry, manual auscultation of the thorax and where necessary, with chest X-ray or CT scan. They wore the WELMO sensors vest for a period of 15-20 minutes during which they performed tidal and deep breathing, cough and spirometry maneuvers and changes of posture. At the end of the study, they were requested to fill in a questionnaire about comfort and usability of the vest.

Patients from various thoracic disease categories were included from both sexes and aged 18-90 years. The study was approved by the bioethics committee of the Hospital and personal data protection provisions were in place. The obtained signals (lung sounds and EIT signals) were examined for consistency with conventionally obtained medical data and the usability, comfort, patient acceptance and practicality of the WELMO vest was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 years
* Suffering from respiratory disease
* Outpatient at Pulmonology Department of G Papanikolaou Hospital
* Hospitalized at Pulmonology Department of G Papanikolaou Hospital
* Hospitalized at 1st ICU of G Papanikolaou Hospital

Exclusion Criteria:

* Age <16 years
* Skin allergies or broken skin
* Unwilling to provide informed consent

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
usability of WELMO vest | 1 day for every patient
  Likert type Questionnaire about the usability /patient acceptance/ ease of wearing/ feeling of restriction of respiration/ aesthetic view of the specialized WELMO sensors vest.

SECONDARY OUTCOMES:
Validity of WELMO vest signals (sounds) | 1 day for every patient
  Comparison of the obtained auscultation signals with conventionally acquired biosignals
Validity of WELMO vest signals (EIT) | 1 day for every patient
  Comparison of the obtained auscultation signals with conventionally acquired biosignals

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Kaimakamis, MD, MSc, PhD, Principal Investigator — 1st ICU, G. papanikolaou Hospital, Thessaloniki, Greece
Locations (1):
- 1st ICU, "G.Papanikolaou" General Hospital of Thessaloniki, Greece, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rocha BM, Filos D, Mendes L, Serbes G, Ulukaya S, Kahya YP, Jakovljevic N, Turukalo TL, Vogiatzis IM, Perantoni E, Kaimakamis E, Natsiavas P, Oliveira A, Jacome C, Marques A, Maglaveras N, Pedro Paiva R, Chouvarda I, de Carvalho P. An open access database for the evaluation of respiratory sound classification algorithms. Physiol Meas. 2019 Mar 22;40(3):035001. doi: 10.1088/1361-6579/ab03ea. PMID 30708353
- [Result] Frerichs I, Vogt B, Wacker J, Paradiso R, Braun F, Rapin M, Caldani L, Chetelat O, Weiler N. Multimodal remote chest monitoring system with wearable sensors: a validation study in healthy subjects. Physiol Meas. 2020 Feb 5;41(1):015006. doi: 10.1088/1361-6579/ab668f. PMID 31891938
- [Result] Frerichs I, Lasarow L, Strodthoff C, Vogt B, Zhao Z, Weiler N. Spatial Ventilation Inhomogeneity Determined by Electrical Impedance Tomography in Patients With Chronic Obstructive Lung Disease. Front Physiol. 2021 Dec 13;12:762791. doi: 10.3389/fphys.2021.762791. eCollection 2021. PMID 34966289
- [Result] Kilintzis V, Alexandropoulos VC, Beredimas N, Maglaveras N. A Methodology for an Auto-Generated and Auto-Maintained HL7 FHIR OWL Ontology for Health Data Management. Stud Health Technol Inform. 2021 Nov 18;287:99-103. doi: 10.3233/SHTI210824. PMID 34795090
- See also: Official website of EU funded WELMO project — http://welmo-project.eu/

DOCUMENTS (1):
  • Study Protocol (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT05531539/Prot_000.pdf